CLINICAL TRIAL: NCT00943293
Title: A Phase I/II Study of Vaccination Against Minor Histocompatibility Antigens HA1 or HA2 After Allogeneic Stem Cell Transplantation for Advanced Hematologic Malignancies
Brief Title: Minor Histocompatibility Vaccination After Allogeneic Stem Cell Transplantation for Advanced Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual; did not enter phase 2
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12175A
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Preleukemia; Myeloproliferative Disorders; Lymphoma; Myeloma; Graft Versus Host Disease
Keywords: GVHD
MeSH Terms: conditions — Preleukemia; Myeloproliferative Disorders; Lymphoma; Neoplasms, Plasma Cell; Graft vs Host Disease | interventions — fludarabine; Melphalan; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental)
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Campath

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2 intravenously daily at the same time over 30 minutes on days -7,-6,-5,4,-3.
Drug: Melphalan — Melphalan 140 mg/m2 IV on day -2.
Drug: Campath — Campath, 20 mg IV on day -7, 6, -5, -4, and -3.

SUMMARY:
This is a clinical research study designed to evaluate whether the administration of a vaccine to patients after transplant consisting of a minor histocompatibility antigen (mHag peptide) mixed with G-CSF (a drug intended to stimulate the immune system) can stimulate increased graft versus leukemia (GVL) responses without causing graft-versus-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory acute myelogenous or lymphoid leukemia.
* Acute myeloid or lymphocytic leukemia in first remission at high-risk for recurrence.
* Chronic myelogenous leukemia in accelerated phase or blast-crisis.
* Chronic myelogenous leukemia in second or subsequent chronic phase
* Recurrent or refractory malignant lymphoma or Hodgkin's disease
* Multiple myeloma at high risk for disease recurrence.
* Chronic lymphocytic leukemia, relapsed or with poor prognostic features.
* Myeloproliferative disorder (polycythemia vera, myelofibrosis) with poor prognostic features.

Exclusion Criteria:

* Clinical progression.
* Contra-indications for vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2003-05; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine in HLA A2 positive patients with hematological malignancies undergoing transplantation from HLA-identical donors, if HA1/2-peptide vaccinations can induce or enhance short- and long-term allogeneic HA1/2-specific T cell immunity. | 5 years

SECONDARY OUTCOMES:
To evaluate if HA1/2 peptide vaccination induces toxicity, especially acute GVHD after HLA-identical transplantation. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Artz, M.D., Principal Investigator — University of Chicago
Locations (1):
- The Uniiversity of Chicago, Chicago, Illinois, United States